CLINICAL TRIAL: NCT04324034
Title: Randomized Study Comparing Endoscopic Transvaginal vNOTES Surgery to Laparoscopy in Terms of Postoperative Pain
Brief Title: vNOTES Transvaginal Endoscopic Surgery Versus Laparoscopy
Acronym: NOTRANDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_1013
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Salpingectomy
Keywords: vNOTES; laparoscopy; salpingectomy; pain
MeSH Terms: conditions — Pain | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vNOTES (Experimental): vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is vaginal surgery with a natural approach. The GelPOINT V-path transvaginal access platform is used. It is a device designed to be placed transvaginally to establish a pathway for the insertion of minimally invasive instruments while maintaining insufflation to perform diagnostic or operative procedures. This device also allows a passage for the extraction of operating parts.
  Interventions: Device: vNOTES
- laparoscopy (Active Comparator): conventional laparoscopy
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Device: vNOTES — vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is vaginal surgery with a natural approach. The GelPOINT V-path transvaginal access platform is used. It is a device designed to be placed transvaginally to establish a pathway for the insertion of minimally invasive instruments while maintaining insufflation to perform diagnostic or operative procedures. This device also allows a passage for the extraction of operating parts.
  Arms: vNOTES
Procedure: laparoscopy — The surgery by conventional laparoscopy is used
  Arms: laparoscopy

SUMMARY:
The feasibility and safety of laparoscopy are no longer to be demonstrated, especially in the field of gynecology, but this technique often causes post-operative pain. New techniques are being developed to overcome the inconvenience of laparoscopy, notably endoscopic transluminal surgery using a natural orifice (NOTES). It avoids incisions and therefore scarring, and could reduce post-operative pain. It is now developing in the field of transvaginal gynecology (vNOTES).

This study is the first prospective randomized study comparing the vNOTES technique to laparoscopy with postoperative pain assessment for performing a salpingectomy. The hypothesis is that the use of vNOTES transvaginal endoscopic surgery would reduce the post-operative pain of patients compared to laparoscopy in the context of a salpingectomy.

ELIGIBILITY:
Inclusion Criteria:

* planned surgery procedure : bilateral salpingectomy for outpatient benign indication
* patients with free, informed and signed consent

Exclusion Criteria:

* disorders leading to an unacceptable risk of postoperative complications sought during the interrogation of the patient (disorders of blood coagulation, disorders of the immune system, progressive diseases ....)
* pregnancy or wish for subsequent pregnancy
* lactating women
* intervention in the context of pelvic cancer
* history of uni- or bilateral salpingectomy
* contraindication to laparoscopy
* history of rectal surgery
* endometriosis
* pelvic inflammatory disease
* genital infection
* not eligible for outpatient care
* associated surgical procedure planned during the intervention (hysterectomy, sub-urethral strip, prolapse cure ...)
* participation in another interventional research related to the gynecological sphere
* inability to understand the information given
* a person not affiliated to a social security scheme, or deprived of liberty, or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Pain score (VAS) | Day 1 (the day after surgery)
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)

SECONDARY OUTCOMES:
Pain score (VAS) | Day 0 (Hour 2 post surgery)
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 100 mm (unbearable pain)
Pain score (VAS) | Day 0 (Hour 6 post surgery)
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 100 mm (unbearable pain)
pain score (VAS) | Day 7
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 100 mm (unbearable pain)
pain score (QDSA) | Day 0 (Hour 6 post surgery)
  Pain score assessed by QDSA short questionnaire (Saint-Antoine Pain Questionnaire) : list of 16 qualifiers to describe pain, score ranging from 0 to 64
pain score (QDSA) | Day 1 (the day after surgery)
  Pain score assessed by QDSA short questionnaire (Saint-Antoine Pain Questionnaire) : list of 16 qualifiers to describe pain, score ranging from 0 to 64
pain score (QDSA) | Day 7
  Pain score assessed by QDSA short questionnaire (Saint-Antoine Pain Questionnaire) : list of 16 qualifiers to describe pain, score ranging from 0 to 64
ease of performing the technique score (VAS) | Day 0 (30 minutes after surgery)
  Visual analogic scale (VAS) is used to evaluate from 0 (very easy) to 100 mm (very difficult).
duration of surgery | Day 0 (30 minutes after surgery)
  duration of surgery (between incision and closure) in minutes
Surgery complications | Month 1
  Description of all per and postoperative complications
outpatient care | Day 1
  number of patients discharged from hospital on the same day of the intervention
dose of morphine | Day 0 (2 hours post surgery)
  total dose of morphine (mg) administered in the post-interventional surveillance room
dose of analgesic | Day 0 (2 hours post surgery)
  total administered dose of analgesic supplement (mg) in post-interventional monitoring room
duration of analgesic | Day 0 (2 hours post surgery)
  duration of analgesic treatment (min) in post-interventional monitoring room
dose of analgesic | Day 0 (8 hours post surgery)
  total administered dose of analgesics (mg) during the hospital stay
duration of analgesic | Day 0 (8 hours post surgery)
  duration of analgesic treatment (hours) during the hospital stay
dose of analgesic | month 1
  total administered dose of analgesics (mg) during the month following the surgery
duration of analgesic | month 1
  duration of analgesic treatment (days) during the month following the surgery
quality of life score | month 1
  assessed by the questionnaire SF-12 (abridged version of the Medical Outcomes Study Short-Form General Health Survey SF-36). It allows to obtain 2 scores: mental and social score (from 5.89058 to 71.966825) and physical score (from 9.94738 to 70.02246). The average of this scores in the general population is 50.
symptom improvement score | month 1
  assessed by the questionnaire PGI-I (Patient Global Impression of Improvement ) (from 1 "much better" to 7 "much worse")
patient satisfaction score | month 1
  Visual analogic scale (VAS) is used to evaluate from 0 (not at all satisfied) to 100 mm (very satisfied).
patient management costs | month 1
  Patient management costs according to the two surgical strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No